CLINICAL TRIAL: NCT06467084
Title: Open-Label Safety, Pharmacokinetic, and Efficacy Trial of Sebetralstat (KVD900) in Pediatric Patients (Ages 2-11) With Hereditary Angioedema Type I or II
Brief Title: Open-Label Safety, PK, and Efficacy Trial of Sebetralstat (KVD900) in Pediatric Patients (Ages 2-11) With HAE Type I or II
Acronym: KONFIDENT-KID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KalVista Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KVD900-303
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hereditary Angioedema
Keywords: KONFIDENT-KID
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — sebetralstat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 150 mg Dose Group (Other): Patients will take a single 150 mg dose of KVD900.
  Interventions: Drug: KVD900 150 mg
- 300 mg Dose Group (Other): Patients will take a single 300 mg dose of KVD900.
  Interventions: Drug: KVD900 300 mg
- 600 mg Dose Group (Other): Patients will take a single 600 mg dose of KVD900.
  Interventions: Drug: KVD900 600 mg

INTERVENTIONS:
Drug: KVD900 150 mg — KVD900 Tablet 150 mg (2 x 75 mg)
  Arms: 150 mg Dose Group
Drug: KVD900 300 mg — KVD900 Tablet 300 mg (1 x 300 mg)
  Arms: 300 mg Dose Group
Drug: KVD900 600 mg — KVD900 Tablet 600 mg (2 x 300 mg)
  Arms: 600 mg Dose Group

SUMMARY:
KVD900-303 is an open-label, multicenter clinical trial in patients aged 2 to 11 years old with HAE Type I or II.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 2 to 11 years of age.
2. Confirmed diagnosis of HAE Type I or II.
3. For patients ≥20 kg at screening, patient has had at least 1 documented HAE attack in the last year prior to screening.
4. Caregiver, as assessed by the Investigator, must be able to appropriately store and administer IMP and be able to read, understand, and complete the diary.
5. Investigator believes that the patient and caregiver are willing and able to adhere to all protocol requirements.
6. Parent or Legally Authorized Representative (LAR) provides signed informed consent and patient provides assent (when applicable).

Exclusion Criteria:

1. Any concomitant diagnosis of another form of chronic angioedema, such as acquired C1 inhibitor deficiency, HAE with normal C1-INH, idiopathic angioedema, or angioedema associated with urticaria.
2. A clinically significant history of poor response to bradykinin receptor 2 blocker, C1-INH therapy, or plasma kallikrein inhibitor therapy for the management of HAE, in the opinion of the Investigator.
3. Patient weighs <9.5 kg.
4. Use of angiotensin-converting enzyme inhibitors after the Screening Visit.
5. Any estrogen-containing medications with systemic absorption (such as oral contraceptives including ethinylestradiol or hormonal replacement therapy) within 7 days prior to the Screening Visit.
6. Patients who require sustained use of strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers or moderate CYP3A4 inducers.
7. Any clinically significant comorbidity or systemic dysfunction, which in the opinion of the Investigator, would jeopardize the safety of the patient by participating in the trial.
8. Known hypersensitivity to sebetralstat or to any of the excipients.
9. Participation in any interventional investigational clinical trial within 4 weeks of the last dosing of investigational drug prior to the Screening Visit.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
The proportion of pediatric patients with HAE Types I or II who take any sebetralstat dose, who experience any AE(s) (including fatal AEs) during the study, irrespective of uses of other medications and sebetralstat discontinuations for any reason. | Throughout the duration of the trial, up to 1 year.

SECONDARY OUTCOMES:
Caregiver Global Impression of Change (CaGI-C): Time to beginning of symptom relief defined as at least "a little better" (2 time points in a row) | Within 12 hours of the first IMP administration.
Caregiver Global Impression of Severity (CaGI-S): Time to first incidence of decrease from baseline (2 time points in a row) | Within 12 hours of the first IMP administration.
CaGI-S: Time to HAE attack resolution defined as "none" | Within 24 hours of the first IMP administration

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — KalVista Pharmaceuticals, Ltd.
Locations (23):
- United States (10):
  - KalVista Investigative Site, Birmingham, Alabama
  - KalVista Investigative Site, Scottsdale, Arizona
  - KalVista Investigative Site, San Diego, California
  - KalVista Investigative Site, Santa Monica, California
  - KalVista Investigative Site, Evansville, Indiana
  - KalVista Investigative Site, Wheaton, Maryland
  - KalVista Investigative Site, St Louis, Missouri
  - KalVista Investigative Site, Toledo, Ohio
  - KalVista Investigative Site, Hershey, Pennsylvania
  - KalVista Investigative Site, Dallas, Texas
- KalVista Investigative Site, Edmonton, Alberta, Canada
- France (3):
  - KalVista Investigative Site, Lille
  - KalVista Investigative Site, Marseille
  - KalVista Investigative Site, Paris
- KalVista Investigative Site, Frankfurt am Main, Germany
- Israel (3):
  - KalVista Investigative Site, Haifa
  - KalVista Investigative Site, Petah Tikva
  - KalVista Investigative Site, Tel Aviv
- Italy (3):
  - KalVista Investigative Site, Milan
  - KalVista Investigative Site, Padua
  - KalVista Investigative Site, Rome
- Japan (2):
  - KalVista Investigative Site, Kawagoe
  - KalVista Investigative Site, Tokyo

IPD SHARING:
Plan to Share IPD: No
Data will not be shared until all global regulatory filings are complete.